CLINICAL TRIAL: NCT05028660
Title: Glycosaminoglycan Profiling for Prognostication of Muscle-invasive Bladder Cancer - a Pilot Study
Brief Title: AURORAX-0093A: Glycosaminoglycan Profiling for Prognostication of Muscle-invasive Bladder Cancer - a Pilot Study
Acronym: AUR93A
Status: Completed | Type: Observational
Sponsor: Elypta (Industry)
Collaborators: Lund University (Other)
Responsible Party: Sponsor
Other Study IDs: ECD-AUR93A001
Record Dates: First submitted 2021-08-25; First posted 2021-08-31 (Actual); Last update posted 2025-05-09 (Actual); Status verified 2025-04

CONDITIONS: Muscle-Invasive Bladder Carcinoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — plasma and urine
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Cohort 1: Sample size of approximately 47 patients with MIBC and elected for NAC
  Interventions: Diagnostic Test: GAG score

INTERVENTIONS:
Diagnostic Test: GAG score — blood and urine samples to determine GAG scores

SUMMARY:
AURORAX-0093A (AUR93A) is a pilot cohort observational study that will explore the use of urine and plasma glycosaminoglycans (GAGs) to prognosticate muscle-invasive bladder cancer (MIBC) patients elected for neo-adjuvant chemotherapy (NAC).

DETAILED DESCRIPTION:
There are around 200 000 cases of bladder cancer (BCa) in the EU every year. Of these, about 25% are diagnosed at a late stage wherein cancer has invaded the muscular wall. The survival of patients with muscle-invasive bladder cancer (MIBC) largely depends on the response to disease management, which in turn is likely dependent on the biology underlying different subtypes of MIBC.

The standard treatment is radical cystectomy (RC) and eligible patients are offered neo-adjuvant chemotherapy (NAC). However, only 30% of these patients report a complete response. Even though the response to NAC is likely correlated to the underlying tumor biology (for example, the TP53-like MIBC subtype is associated with a higher frequency of resistance to NAC), there are today no approved biomarkers to select patients likely to benefit from NAC. This information could in turn translate into more precise and personalized treatment for the patient.

In a proof-of-concept prospective study, we discovered that the profiling of urine and plasma glycosaminoglycans (GAGs) could be useful for the diagnosis and prognosis of BCa. AUR93A is a prospective single-arm cohort exploratory study. A sample size of approx. 47 patients with MIBC and elected for NAC will be included in this study and it is assumed that 30% will experience complete response at the post-operative visit. The goal is to correlate baseline (pre-NAC) GAGs to complete response rate (CRR) after RC and recurrence-free survival (RFS).

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of transitional cell carcinoma of the bladder (mixed histology tumors allowed if transitional cell histology is predominant [50%+] histology)
* Clinical stage T2-T4a N0-N2 M0 by CT (or MRI) + PET/CT
* Elected and fit according to institutional guidelines for cisplatin-based NAC followed by RC
* ECOG score 0-1

Exclusion Criteria:

* Previously intravenous chemotherapy for bladder cancer. (Patients who have had previous radiotherapy or concurrent chemo-radiation for bladder cancer are still eligible.)
* Currently participating or has participated in a study of an investigational agent and received study therapy or received investigational device within 4 weeks before the first dose NAC
* Known additional malignancy that is progressing or requires active treatment except for basal cell carcinoma of the skin, or squamous cell carcinoma of the skin that has undergone potentially curative therapy, or in situ cervical cancer.

(A history of prostate cancer that was treated with definitive intent (surgically or through radiation therapy) is acceptable provided that the following criteria are met: Stage T2N0M0 or lower, Gleason score less/equal to 7 and prostatic-specific antigen (PSA) undetectable for at least 1 year while off androgen deprivation therapy that was either treated with definitive intent or untreated in active surveillance that has been stable for the past year before study allocation. Pathological evidence of concurrent T1a/b prostate cancer after radical cystecto-prostatectomy are still eligible.)

- Evidence of measurable nodal or metastatic disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will enroll patients with MIBC elected for NAC, defined as:
  * MIBC: pathologically confirmed transitional cell carcinoma of the bladder with the invasion of the bladder muscular wall and no evidence of regional or distal metastases (T2-T4a cN0-N2 M0)
  * NAC: any choice of cisplatin-containing chemotherapeutic regimen.
Sampling Method: Probability Sample
Enrollment: 43 (Actual)
Dates: Start 2021-07-21 (Actual); Primary Completion 2025-04-30 (Actual); Study Completion 2025-04-30 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with complete response at the post-operative visit after RC. | 15 to 90 days after radical cystectomy surgery
  Percentage point difference in complete response rates between GAG favorable and GAG poor patients

SECONDARY OUTCOMES:
Proportion of patients with recurrence at any time after treatment | 15 to 90 days after radical cystectomy surgery
  Percentage point difference in recurrence rates between GAG favorable and GAG poor patients
Proportion of complete responses after NAC according to CT-based RECIST v1.1 | 15 to 90 days after radical cystectomy surgery
  Percentage point difference in complete response rates after NAC between GAG favorable and GAG poor patients

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Gatto, Study Director — Elypta, Solna, Sweden
Locations (5):
- Zealand University Hospital, Roskilde, Denmark
- Italy (3):
  - AOU Careggi, Florence
  - IRCCS Ospedale San Raffaele, San Raffaele Hospital, Milan
  - IRCCS Regina Elena, Rome
- Sahlgrenska University Hospital, Gothenburg, Sweden

IPD SHARING:
Plan to Share IPD: Undecided
Unidentified clinical and biochemical data will become available to the research community along with the publication of a scientific article related to the present investigation.